CLINICAL TRIAL: NCT05986981
Title: Single-arm, Open-label Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of MUC1 Therapeutic Tumor Vaccine in Advanced Solid Cancers
Brief Title: MUC1 Therapeutic Tumor Vaccine in Advanced Solid Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCHVaccineMUC1
Record Dates: First submitted 2023-05-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor, Adult
Keywords: vaccine; Mucin 1; MUC1; malignant tumor
MeSH Terms: conditions — Medullary cystic kidney disease 1; Neoplasms | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: The study flow included a screening period (week -4 to day -1), a treatment period (day 1 to week 8 or 16, including a DLT observation period on days 1-28), an end-of-treatment visit, and a survival follow-up. The treatment period included the initial treatment period (day 1 to week 8) and the augmentation period (week 12 to week 16). Subjects after signing and providing formal informed consent entered the screening period, during which eight separate administrations of the vaccine were administered, of which the investigator determined whether to continue treatment from week 8 to week 12 based on a combination of efficacy, safety, and adherence.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MUC1 Vaccine (Experimental): Enrollment by cohort from the starting dose of the trial and proceed to the next higher dose level if no one of the first 3 subjects develops DLT. If 1 of the 3 subjects develops DLT, then 3 additional subjects will be added to that dose level for a total of 6 subjects.
  If only 1 of 6 subjects develops DLT, proceed to the next higher dose level. If no fewer than 2 of the 6 subjects develop DLT, no more subjects will be added to that dose level and dose escalation will cease. The Safety Monitoring Committee (SMC) decides whether to use the intermediate dose as the next dose level for the study. Until the maximum sample size specified in the protocol or the SMC decides to terminate the dose increment.each subject receives only one dose group of study drug (during the incremental period, subjects may receive a reduced dose to continue treatment after the investigator has assessed the risk-benefit for safety reasons; dose increments are not permitted for the same subject).
  Interventions: Drug: Vaccine

INTERVENTIONS:
Drug: Vaccine — Dose-escalation trial, according to the classic "3+3" model, divided into three dose levels of 0.5 mg, 1.0 mg, 2.0 mg for enrollment, is expected to enroll a total of 9-18 subjects (0.5 mg dose group to be enrolled in 3-6 subjects, 1.0 mg dose group is proposed to be enrolled in 3-6 subjects, 2.0 mg dose group is proposed to be enrolled in 3-6 subjects, and the dose group is proposed to be enrolled in 3-6 subjects, and the dose group is proposed to be enrolled in 3-6 subjects. dose group is proposed to include 3-6 subjects).

SUMMARY:
This is an investigator-initiated, single-center, open, single-arm, exploratory study of a therapeutic cancer vaccine for the treatment of advanced solid tumors. A dose-escalation trial is being conducted in subjects diagnosed with advanced solid tumors to evaluate the safety and tolerability of the cancer vaccine in subjects with advanced solid tumors and to preliminarily evaluate the efficacy of the tumor vaccine in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Malignant tumours have become one of the major public health problems that seriously threaten human health. According to the latest global cancer burden data for 2020 released by the International Agency for Research on Cancer (IARC) of the World Health Organization (WHO), there will be 19.29 million new cancer cases and 9.96 million deaths globally in 2020; in 2020, there will be 4.57 million new cancer cases and 3 million deaths in China, with the number of new cancers in China accounting for 23.7% of the global incidence and 30% of the global deaths, both of which are the highest in the world. The number of new cancer cases in China accounts for 23.7% of global incidence and the number of cancer deaths accounts for 30% of global deaths, both of which rank first in the world, with lung, liver, stomach, esophagus and colorectal cancers having the highest mortality rates.

At present, in addition to the traditional surgery, radiotherapy and chemotherapy treatments for malignant tumours, with the advancement of biological sciences, tumour immunotherapy has developed significantly, in which antibody drugs and cell therapy (chimeric antigen receptor T cell, CAR-T) have products on the market. With the deepening research on the characteristics of tumour cells and the differences in protein expression, therapeutic cancer vaccines have gradually moved from theory to practice and have shown good performance in clinical trials.

The therapeutic cancer vaccine YB-01 is a therapeutic cancer vaccine formulation developed by the Department of Nuclear Medicine of Peking Union Medical College Hospital and commissioned to be produced by Zhaoyan Biologicals, a company with the qualification of Good manufacturing practice (GMP), and developed by Yuanben (Zhuhai Hengqin) Biotech Co. YB-01 cancer vaccine is a recombinant fusion protein with aluminium adjuvant and CpG182 adjuvant, and its core component is Mucin N-terminal region (MNR), which is specifically expressed by cancer cells. Mucin1 (MUC1) is a glycoprotein that plays a pivotal role in tumour formation, growth, invasion, signalling, pro-angiogenesis, anoxia and chemoresistance. Normal epithelial cells exist with low expression of MUC1, whereas cancerous cells have high expression of MUC1 (100-fold increase), and this differential expression is due to the fact that it is abnormally pronounced in biliary pancreatic carcinoma, cholangiocarcinoma, gastric adenocarcinoma, breast carcinoma and neuroendocrine pancreatic carcinoma, so that vaccine-induced immune response is only directed against the cancerous cells, but not against the normal tissues, and non-glycosylated MUC1 has become an important target for cancer therapy.YB- 01 vaccine targets MUC1 and enhances humoral and cell-mediated immune responses through immunity to MUC1 peptide or MUC1 peptide-activated dendritic cells (DC).DC cells activate CD4 T cells, which promotes the activation of B cells to produce antibodies against MUC1, and DC cells also activate CD8 T cells, which target and kill tumour cells that express MUC1. cells expressing MUC1.

Approximately 9-18 subjects will be recruited in this study. The investigational drug used in the study is the therapeutic cancer vaccine YB-01, and the study is designed to investigate the safety, tolerability, and preliminary efficacy of the vaccine in subjects with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

1. screening period patients are able to understand and voluntarily sign an informed consent form;
2. males and females between the ages of 18 and 75 years (both ends included);
3. expected survival ≥ 3 months;
4. advanced subjects with histologically or cytologically proven advanced solid tumors who have failed standard multiline therapy;
5. have at least one measurable lesion (i.e., mass ≥10 mm in diameter and malignant lymph node ≥15 mm in short diameter on enhanced scan with layer thickness ≤5 mm on spiral CT) according to the efficacy evaluation criteria for solid tumors, RECIST version 1.1 (see Appendix 4, Criteria for Evaluating the Efficacy of Solid Tumor Treatments);
6. Fresh or archived tumor tissue samples within 5 years are available for central laboratory testing during the screening period (if they are truly unavailable, this will not affect enrollment);
7. ECOG physical status score of 0 to 2;
8. treatment with other anti-tumor drugs (e.g., chemotherapy, hormone therapy, immunotherapy, antibody therapy, radiotherapy) prior to the first dose exceeds the 5 half-life of the drug or more than 4 weeks before the first dose (whichever is shorter);
9. Organ function levels must meet the following requirements (no blood or blood product transfusion, hematopoietic stimulating factor, albumin, or blood product use within 14 days prior to the examination): absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count (PLT) ≥ 75 × 109/L, hemoglobin (Hb) ≥ 90 g/L; serum total bilirubin (TBIL) ≤ 1.5 Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value, glutamic transaminase (AST) and alanine aminotransferase (ALT) ≤2.5 times the upper limit of normal value (if liver metastasis is present, total bilirubin ≤3 times the upper limit of normal value, AST and ALT ≤5 times the upper limit of normal value are allowed). 10;
10. Pre-menopausal women of childbearing potential must undergo a pregnancy test within 7 days prior to the start of treatment, and the result of the pregnancy test must be negative and non-lactating; women without childbearing potential may not undergo a pregnancy test and contraception, provided they are over 50 years of age, have not used hormone therapy and have stopped menstruating for at least 12 months, or have been sterilized. All enrolled subjects (either male or female) should use adequate barrier contraception throughout the treatment period and for 3 months after completion of treatment.
11. Other toxicity parameters must be NCI-CTCAE v.5.0 Grade 0 or 1.

Exclusion Criteria:

1. Subjects who require long-term systemic application of anti-allergic medications or who have a history of life-threatening allergic reactions to any vaccine or medication;
2. those with symptomatic or rapidly progressing central system metastases. Presence of extensive pulmonary metastases causing respiratory distress; subjects with tumours in close proximity to or invading large blood vessels or nerves;
3. new cerebrovascular accidents (including ischaemic stroke, haemorrhagic stroke and transient ischaemic attack) within 6 months prior to screening;
4. acute myocardial infarction, uncontrolled angina pectoris, uncontrolled arrhythmia, severe heart failure (see Appendix 3, New York Heart Association's Heart Failure Classification Criteria, NYHA Class ≥ III) and other cardiovascular diseases within 6 months prior to screening;
5. have received immunomodulatory medications within 4 weeks prior to the date of first vaccination (D1), including, but not limited to, IL-2, CTLA-4 inhibitors, CD40 agonists, CD137 agonists, and IFN-alpha (except for high-risk surgical subjects using IFN-alpha as an adjuvant therapy if IFN-alpha therapy was discontinued within the 4 weeks prior to the date of the trial);
6. those with a history of renal insufficiency with serum creatinine levels greater than 1.5 times the upper limit of normal;
7. have received a blood transfusion, erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), or granulocyte-macrophage colony-stimulating factor (GM-CSF) within 2 weeks prior to the first dose of drug;
8. subjects with skin conditions that may prevent intradermal vaccine from reaching the target area (e.g., psoriasis);
9. subjects in the Screening Period who continue to have adverse reactions from prior anti-neoplastic therapy that have not been restored to a CTCAE Version 5.0 grade rating of ≤ Grade 1 (with the exception of alopecia and platinum-induced neurotoxicity of ≤ Grade 2);
10. need for concomitant use of steroidal hormonal medications (tumour or non-tumour related disease); exceptions may be made for those requiring topical (not applied to the vaccination site) or inhaled steroids;
11. the presence of active or uncontrollable infections requiring systemic therapy (except for simple urinary tract infections or upper respiratory tract infections) in the subject within 4 weeks prior to screening; and the presence of antibodies to the Human Immunodeficiency Virus (HIV), hepatitis B Surface Antigen (SAB) positive and/or hepatitis B Core Antibody (HBCO) positive with Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) >1000 copies/mL and Hepatitis C virus (HCV) antibodies on virological testing during the Screening Period, Subjects who are positive for antibodies specific to syphilis spirochetes;
12. poorly controlled hypertension (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) after treatment;
13. subjects with a history of autoimmune disease [e.g., the following, but not limited to: interstitial pneumonitis, uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism (hypothyroidism without clinical symptoms or hypothyroidism due to radiotherapy may be included), subjects with vitiligo or cured asthma that does not currently require any intervention may be included, subjects requiring bronchodilators for medical intervention cannot be included];
14. subjects with active ulcers or gastrointestinal bleeding during the Screening Period;
15. subjects who have received a previous similar therapeutic cancer vaccine or who have received another vaccine within 4 weeks prior to Screening;
16. subjects with congenital or acquired immunodeficiency;
17. subjects who have participated in other clinical trials within 1 month prior to screening;
18. subjects with known alcohol or drug addiction;
19. subjects who, in the opinion of the investigator, have an underlying health condition, mental condition, or social condition that makes the subject unable or unwilling to comply with the study protocol
20. any other condition which, in the opinion of the Investigator, makes participation in this study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The safety of the vaccine using CTCAE v5.0 based on the number of patients with treatment-related adverse events. | 8~12weeks
  Assess the safety of the vaccine using CTCAE v5.0 based on the number of patients with treatment-related adverse events.
DLT | 8~12weeks
  Inject 0.5 to 2.0 mg of vaccine intramuscularly over a 16-week cycle to determine dose-limiting toxicity (DLT).
RP2D | 8~12weeks
  Determine if the maximum tolerated dose is among the doses explored and determine the recommended phase 2 dose (RP2D) of the vaccine.

SECONDARY OUTCOMES:
Preliminary assessment of the effectiveness of therapeutic oncology vaccines in advanced solid tumors. | 2years
  Preliminary assessment of the effectiveness of therapeutic oncology vaccines in advanced solid tumors.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold M, Morgan E, Rumgay H, Mafra A, Singh D, Laversanne M, Vignat J, Gralow JR, Cardoso F, Siesling S, Soerjomataram I. Current and future burden of breast cancer: Global statistics for 2020 and 2040. Breast. 2022 Dec;66:15-23. doi: 10.1016/j.breast.2022.08.010. Epub 2022 Sep 2. PMID 36084384
- [Background] Rumgay H, Shield K, Charvat H, Ferrari P, Sornpaisarn B, Obot I, Islami F, Lemmens VEPP, Rehm J, Soerjomataram I. Global burden of cancer in 2020 attributable to alcohol consumption: a population-based study. Lancet Oncol. 2021 Aug;22(8):1071-1080. doi: 10.1016/S1470-2045(21)00279-5. PMID 34270924
- [Background] O'Donnell JS, Teng MWL, Smyth MJ. Cancer immunoediting and resistance to T cell-based immunotherapy. Nat Rev Clin Oncol. 2019 Mar;16(3):151-167. doi: 10.1038/s41571-018-0142-8. PMID 30523282
- [Background] Lei K, Kurum A, Kaynak M, Bonati L, Han Y, Cencen V, Gao M, Xie YQ, Guo Y, Hannebelle MTM, Wu Y, Zhou G, Guo M, Fantner GE, Sakar MS, Tang L. Cancer-cell stiffening via cholesterol depletion enhances adoptive T-cell immunotherapy. Nat Biomed Eng. 2021 Dec;5(12):1411-1425. doi: 10.1038/s41551-021-00826-6. Epub 2021 Dec 6. PMID 34873307
- [Background] Riley RS, June CH, Langer R, Mitchell MJ. Delivery technologies for cancer immunotherapy. Nat Rev Drug Discov. 2019 Mar;18(3):175-196. doi: 10.1038/s41573-018-0006-z. PMID 30622344
- [Background] Szeto GL, Finley SD. Integrative Approaches to Cancer Immunotherapy. Trends Cancer. 2019 Jul;5(7):400-410. doi: 10.1016/j.trecan.2019.05.010. PMID 31311655
- [Background] Zhang Y, Zhang Z. The history and advances in cancer immunotherapy: understanding the characteristics of tumor-infiltrating immune cells and their therapeutic implications. Cell Mol Immunol. 2020 Aug;17(8):807-821. doi: 10.1038/s41423-020-0488-6. Epub 2020 Jul 1. PMID 32612154
- [Background] Gao T, Cen Q, Lei H. A review on development of MUC1-based cancer vaccine. Biomed Pharmacother. 2020 Dec;132:110888. doi: 10.1016/j.biopha.2020.110888. Epub 2020 Oct 21. PMID 33113416
- [Background] Nabavinia MS, Gholoobi A, Charbgoo F, Nabavinia M, Ramezani M, Abnous K. Anti-MUC1 aptamer: A potential opportunity for cancer treatment. Med Res Rev. 2017 Nov;37(6):1518-1539. doi: 10.1002/med.21462. Epub 2017 Jul 31. PMID 28759115
- [Background] Hossain MK, Wall KA. Immunological Evaluation of Recent MUC1 Glycopeptide Cancer Vaccines. Vaccines (Basel). 2016 Jul 26;4(3):25. doi: 10.3390/vaccines4030025. PMID 27472370
- [Background] Park JA, Park S, Park HB, Han MK, Lee Y. MUC1-C Contributes to the Maintenance of Human Embryonic Stem Cells and Promotes Somatic Cell Reprogramming. Stem Cells Dev. 2021 Nov 1;30(21):1082-1091. doi: 10.1089/scd.2021.0185. Epub 2021 Oct 18. PMID 34514853
- [Background] Rajabi H, Kufe D. MUC1-C Oncoprotein Integrates a Program of EMT, Epigenetic Reprogramming and Immune Evasion in Human Carcinomas. Biochim Biophys Acta Rev Cancer. 2017 Aug;1868(1):117-122. doi: 10.1016/j.bbcan.2017.03.003. Epub 2017 Mar 14. PMID 28302417
- [Background] Nath S, Mukherjee P. MUC1: a multifaceted oncoprotein with a key role in cancer progression. Trends Mol Med. 2014 Jun;20(6):332-42. doi: 10.1016/j.molmed.2014.02.007. Epub 2014 Mar 22. PMID 24667139
- [Background] Chen W, Zhang Z, Zhang S, Zhu P, Ko JK, Yung KK. MUC1: Structure, Function, and Clinic Application in Epithelial Cancers. Int J Mol Sci. 2021 Jun 18;22(12):6567. doi: 10.3390/ijms22126567. PMID 34207342
- [Background] Macao B, Johansson DG, Hansson GC, Hard T. Autoproteolysis coupled to protein folding in the SEA domain of the membrane-bound MUC1 mucin. Nat Struct Mol Biol. 2006 Jan;13(1):71-6. doi: 10.1038/nsmb1035. Epub 2005 Dec 20. PMID 16369486
- [Background] Raina D, Kharbanda S, Kufe D. The MUC1 oncoprotein activates the anti-apoptotic phosphoinositide 3-kinase/Akt and Bcl-xL pathways in rat 3Y1 fibroblasts. J Biol Chem. 2004 May 14;279(20):20607-12. doi: 10.1074/jbc.M310538200. Epub 2004 Mar 3. PMID 14999001
- [Background] Ota S, Miyashita M, Yamagishi Y, Ogasawara M. Baseline immunity predicts prognosis of pancreatic cancer patients treated with WT1 and/or MUC1 peptide-loaded dendritic cell vaccination and a standard chemotherapy. Hum Vaccin Immunother. 2021 Dec 2;17(12):5563-5572. doi: 10.1080/21645515.2021.2003645. Epub 2021 Dec 17. PMID 34919493